CLINICAL TRIAL: NCT00810836
Title: A Phase 2a, Randomised, Double-Blind, Placebo-Controlled, Multicentre Study to Evaluate the Efficacy, Safety and Tolerability of BG00012 When Given With Methotrexate to Subjects With Active RA Who Have Had an Inadequate Response to Conventional Disease-Modifying Anti-rheumatic Drug Therapy
Brief Title: Efficacy and Safety Study of BG00012 With Methotrexate in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec,Immunology department, Biogen Idec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 109RA201
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): BG00012 480 mg/day
  Interventions: Drug: BG00012
- 2 (Active Comparator): BG00012 720 mg/day
  Interventions: Drug: BG00012
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: BG00012 — oral
  Arms: 1
Drug: BG00012 — Oral
  Arms: 2
Drug: placebo — oral placebo
  Arms: 3

SUMMARY:
The purpose of this study is to investigate whether the drug BG00012 can improve the symptoms of rheumatoid arthritis (RA) in patients who are already taking methotrexate for RA, but who still suffer symptoms of RA. The purpose is also to ensure that the combination of methotrexate is safe for patients to take and that any side effects are acceptable to patients with RA.

DETAILED DESCRIPTION:
The study is a double-blind, placebo-controlled study of BG00012 plus methotrexate, versus methotrexate alone, in patients with active RA, who have had an incomplete response to other conventional disease modifying anti-rheumatic (DMARD) therapy.

ELIGIBILITY:
Inclusion Criteria:

* must be taking methotrexate
* inadequate response to at least one conventional DMARD
* swollen and tender joint count

Exclusion Criteria:

* previous treatment with TNF or any other biologic or prosorba column

Other criteria also apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is the proportion of subjects with ACR20 response in their RA at Week 12. | 12 weeks

SECONDARY OUTCOMES:
To determine the safety and tolerability of BG00012 with methotrexate in this population. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (24):
- Australia (2):
  - Research Site, Woolloongabba, Queensland
  - Research Site, Woodville, South Australia
- Canada (4):
  - Research Site, Sarnia, Ontario
  - Research Site, New Market
  - Research Site, Ottawa
  - Research Site, Rothesay
- Czechia (4):
  - Research Site, Active, Not Recruiting
  - Research Site, Pardubice
  - Research Site, Uh. Hradiste
  - Research Site, Zlín
- India (4):
  - Research Site, Bangalore
  - Research Site, Hyderabaad
  - Research Site, Hyderabad
  - Research Site, Lucknow
- Poland (6):
  - Research Site, Bialystock
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Torun
  - Research Site, Warsaw
- Slovakia (4):
  - Research Site, Banska Bysterica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Piešťany